CLINICAL TRIAL: NCT03644056
Title: A Phase 1, Open-label, Multiple-ascending Dose Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of IMC-001 in Subjects With Metastatic or Locally-advanced Solid Tumors
Brief Title: Dose-escalation Study of IMC-001 in Subject With Metastatic or Locally-advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmuneOncia Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMC-001-101
Record Dates: First submitted 2018-08-17; First posted 2018-08-23 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Solid Tumor; Metastasis; Locally Advanced
Keywords: IMC-001
MeSH Terms: conditions — Neoplasm Metastasis | interventions — IMC-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMC-001 (Experimental): Multiple Dose Level (IMC-001 2 mg/kg etc. every 2 weeks)
  Interventions: Drug: IMC-001

INTERVENTIONS:
Drug: IMC-001 — Different IMC-001 dose level for each cohort group (IMC-001 2 mg/kg etc. every 2 weeks)
  Other Names: Not confirm yet

SUMMARY:
This is a phase 1, Open-label, Multiple-ascending Dose Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of IMC-001 in Subjects with Metastatic or Locally-advanced Solid Tumors

DETAILED DESCRIPTION:
IMC-001 is a PD-L1 targeting, fully human monoclonal antibody. The purpose of this study is to determine safety and evaluate PK, PD and clinical activity of IMC-001. Multiple dose levels of IMC-001 will be tested in subjects with metastatic or locally-advanced solid tumors. Data from this study will also help determine the recommended phase 2 dose of IMC-001.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF).
2. Adult (19 years or older).
3. Histologically or cytologically proven metastatic or locally-advanced solid tumors

Exclusion Criteria:

1. Treatment with non-permitted drugs (within the past 28 days of Screening), including but not limited to systemic immunosuppressive agents, any other investigational medicinal product (IMP), anti-coagulant, or live vaccines.
2. Any prior cancer immunotherapy
3. Concurrent anticancer treatments

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Occurrence of DLTs | During the first 21 days of treatment
  To investigate the occurrence of DLTs of IMC-001 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Jeong Song, CMO/CEO, Study Director — ImmuneOncia Therapeutics Inc.
Locations (1):
- ImmuneOncia, Yongin-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Keam B, Ock CY, Kim TM, Oh DY, Kang WK, Park YH, Lee J, Lee JH, Ahn YH, Kim HJ, Chang SK, Park J, Choi JY, Song YJ, Park YS. A phase I study of IMC-001, a PD-L1 blocker, in patients with metastatic or locally advanced solid tumors. Invest New Drugs. 2021 Dec;39(6):1624-1632. doi: 10.1007/s10637-021-01078-6. Epub 2021 Jul 16. PMID 34268711